CLINICAL TRIAL: NCT00002071
Title: A Double-Blind, Placebo-Controlled Study With Open-Label Follow-Up To Determine the Safety and Efficacy of r-HuEPO in AIDS Patients With Anemia Induced by Their Disease and AZT Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ortho Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 004A; 87-020
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-12

CONDITIONS: HIV Infections; Cytopenias
Keywords: Recombinant Proteins; Erythropoietin; Acquired Immunodeficiency Syndrome; Anemia; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Acquired Immunodeficiency Syndrome; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
To determine the safety and efficacy of erythropoietin administered to AIDS patients with anemia secondary to their disease and/or concomitant zidovudine (AZT) therapy.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* History of any primary hematologic disease.
* Clinically significant disease / dysfunction of the pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems not attributable to underlying AIDS.
* AIDS-related dementia.
* Uncontrolled hypertension (diastolic blood pressure 100 mmHg).
* Presence of concomitant iron deficiency.
* Anemia attributable to factors other than AIDS or zidovudine (AZT) therapy.
* Acute opportunistic infection.
* History of seizures.

Patients with clinically significant disease / dysfunction of the pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems not attributable to underlying AIDS are excluded.

Prior Medication:

Excluded within 30 days of study entry:

* Experimental drug or experimental device.
* Cytotoxic chemotherapy.
* Excluded within 2 months of study entry:
* Androgen therapy.

Clinical diagnosis of AIDS related anemia.

* Clinical diagnosis of AIDS.
* Clinically stable for 1 month preceding study entry.

Substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ortho Pharmaceutical Corp, Raritan, New Jersey, United States

REFERENCES:
- [Background] Rarick M, Wilson E, Bernstein-Singer M, Gill PS, Muggia F, Levine AM. Double-blind placebo controlled study of recombinant human erythropoietin in AIDS patients with anemia caused by HIV infection and zidovudine. Int Conf AIDS. 1989 Jun 4-9;5:195 (abstract no MBO48)